CLINICAL TRIAL: NCT03958656
Title: A Phase I Clinical Trial of T-cells Expressing an Anti-SLAMF7 CAR for Treating Multiple Myeloma
Brief Title: T-cells Expressing an Anti-SLAMF7 CAR for Treating Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, James Kochenderfer, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 190102; 19-C-0102
Record Dates: First submitted 2019-05-21; First posted 2019-05-22 (Actual); Results first posted 2021-09-09 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-08

CONDITIONS: Myeloma-Multiple; Myeloma, Plasma-Cell
Keywords: Chimeric Antigen Receptors; B-cell Maturation Antigen; Immunotherapy; Adoptive T Cell Therapy
MeSH Terms: conditions — Multiple Myeloma | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate; AP 1903 reagent; SLAMF7 protein, human; Receptors, Chimeric Antigen; Automobiles

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/Conditioning Chemotherapy Plus Chimeric Antigen Receptor (CAR) T-cells Dose Escalation (Experimental): Patients will receive escalating doses (up to 4 planned) of Anti-Signaling lymphocytic activation molecule F7 (SLAMF7)-CAR+ T cells infused on day 0 + Cyclophosphamide: 300 mg/m^2 intravenous (IV) infusion over 30 minutes on days -5, -4 and -3 + Fludarabine: 30 mg/m^22 IV infusion over 30 minutes administered immediately following the cyclophosphamide on days -5, -4, and -3
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Rimiducid; Biological: Anti-Signaling lymphocytic activation molecule F7 (SLAMF7) chimeric antigen receptor (CAR) T cells
- 2/Conditioning Chemotherapy Plus Chimeric Antigen Receptor (CAR) T-cells Expansion Phase (Experimental): Maximum tolerated dose (MTD) dose of Anti-Anti-Signaling lymphocytic activation molecule F7 (SLAMF7)- CAR T Cells + Cyclophosphamide: 300 mg/m^2 intravenous (IV) infusion over 30 minutes on days -5, -4 and -3 + Fludarabine: 30mg/m^2 IV infusion over 30 minutes administered immediately following the cyclophosphamide on days -5, -4, and -3
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Rimiducid; Biological: Anti-Signaling lymphocytic activation molecule F7 (SLAMF7) chimeric antigen receptor (CAR) T cells

INTERVENTIONS:
Drug: Cyclophosphamide — 300 mg/m^2 intravenous (IV) over 30 minutes on days -5, -4, and -3
  Other Names: Cytoxan
Drug: Fludarabine — 30 mg/m^2 intravenous (IV) over 30 minutes immediately following the cyclophosphamide on day -5, -4, and -3
  Other Names: Fludara
Drug: Rimiducid — 0.4 mg/kg of Rimiducid intravenous (IV) over 2 hours. (A maximum of 2 doses separated by at least 48 hours) Note: Rimiducid may be administered as needed based on the patient condition at the discretion of the Principal Investigator.
  Other Names: AP1903
Biological: Anti-Signaling lymphocytic activation molecule F7 (SLAMF7) chimeric antigen receptor (CAR) T cells — 0.3x10^6- 12.0x10^6 CAR+ T cells per kg of recipient bodyweight one-time dose on day 0

SUMMARY:
Background:

Multiple myeloma is a blood cancer that is usually incurable. T cells are part of the immune system. Researchers think changing a person's T cells to recognize their cancer could help the person's body kill tumor cells. This is a new approach that uses a patient's own cells to target multiple myeloma.

Objective:

To see if giving anti-Signaling lymphocytic activation molecule F7 (SLAM7) chimeric antigen receptor (CAR) T cells with a stop switch to people with multiple myeloma is safe and to see if adding a gene to stop T-cell activity can limit toxicity of this therapy.

Eligibility:

People ages 18-73 with multiple myeloma for which prior standard treatment has not worked

Design:

Participants will be screened with:

* Medical history
* Physical exam
* Blood, urine, and heart tests
* Bone marrow samples: A needle inserted into the participant's bone will remove marrow.
* Imaging scans: Participants will lie in a machine that takes pictures of the body.

Participants will have apheresis. They will receive a catheter or central line: A plastic tube will be inserted into a chest or arm vein. Blood will be removed and the T cells separated. The rest of the blood will be returned to the participant. The T cells will be manipulated in the lab.

Participants will get chemotherapy through the central line for 3 days.

Participants will receive the manipulated T cells through the central line. They will stay in the hospital at least 9 days.

Participants will have follow-up visits 2 weeks then 1, 2, 3, 4, 6, 9, and 12 months after the infusion. They will then have visits every 6 months for 3 years. Then they will be contacted once per year for 15 years. All visits will include blood tests, and 3 visits will include bone marrow biopsies....

DETAILED DESCRIPTION:
Background:

* Multiple myeloma (MM) is a nearly always incurable malignancy of plasma cells.
* T cells can be genetically modified to express chimeric antigen receptors (CARs) that target malignancy-associated antigens.
* Signaling lymphocytic activation molecule F7 (SLAM7) is highly and uniformly expressed on MM cells but is absent on normal tissues except for some leukocytes, including a subset of cluster of differentiation 8 (CD8)+ T cells, natural killer (NK) cells, B cells, plasma cells and monocytes.
* We have constructed a novel anti-SLAMF7 CAR that can specifically recognize SLAMF7- expressing target cells and eradicate SLAMF7-expressing tumors in mice.
* This protocol will test genetic modification of autologous T cells with genes encoding an inducible caspase 9 (IC9) cell-suicide system plus the anti-SLAMF7 CAR.
* Administration of the dimerizer drug Rimiducid (AP1903) is necessary to activate the inducible caspase 9 (IC9) suicide gene and eliminate CAR T cells.
* In this protocol, the suicide gene system will be used to eliminate CAR-expressing T cells in case of severe toxicities caused by the CAR T cells.
* Possible toxicities include cytokine-associated toxicities such as hypotension, and neurological toxicities. Elimination of NK cells and normal plasma cells could make patients more susceptible to infections. Unknown toxicities are also possible.

Objectives:

Primary

- Determine the safety, feasibility of administering T cells expressing an anti-SLAMF7 CAR plus IC9 cell-suicide system to patients with MM.

Eligibility:

* Greater than or equal to 18 years of age and less than or equal to age 73.
* Patients must have measurable MM defined as a serum M-protein >=0.6 g/dL or a urine M-protein >=200 mg/24 hours or an involved serum free light chain (FLC) level >=10 mg/dL (provided FLC ratio is abnormal) or a biopsy-proven plasmacytoma of 1.5 cm or more in largest dimension, or greater than or equal to 30% bone marrow plasma cells.
* Patients must have previously received at least 3 different treatment regimens for MM.
* Patients must have prior exposure to an immunomodulatory drug (IMiD) such as lenalidomide, and a proteasome inhibitor
* Patients must have a creatinine level of less than or equal to 1.5 mg/dL
* Patients must have a cardiac ejection fraction >= 50%.
* An Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 is required.
* Patients on any anticoagulant medications except aspirin are not eligible.
* No active infections are allowed.
* Absolute neutrophil count >= 1000/microL, platelet count >= 55,000/microL, hemoglobin >= 8g/dL
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less than or equal to 2.5-fold higher than the upper limit of normal.
* At least 14 days must elapse between the time of any prior systemic treatment (including corticosteroids) and the required leukapheresis.
* At least 14 days must elapse between the time of any prior systemic treatment and initiation of protocol treatment. Systemic therapy includes corticosteroids at a dose equivalent to more than 5 mg of prednisone.
* Bone marrow plasma cells must make up less than or equal to 50% of total bone marrow cells less than or equal to 24 days prior to the start of protocol treatment.
* The patient's MM will need to be assessed for SLAMF7 expression by flow cytometry or immunohistochemistry performed at the National Institutes of Health (NIH). The myeloma must express SLAMF7. If unstained, paraffin-embedded bone marrow or plasmacytoma sections are available from prior biopsies, these can be used to determine SLAMF7 expression by immunohistochemistry; otherwise patients will need to come to the NIH for a bone marrow biopsy or other biopsy of a plasmacytoma to determine SLAMF7 expression. The sample for SLAMF7 expression can come from a biopsy obtained at any time before enrollment.

Design:

* This is a phase I dose-escalation trial
* Patients will undergo leukapheresis, and T cells will be modified to express the IC9-anti-SLAMF7 CAR construct.
* The chemotherapy conditioning regimen is cyclophosphamide 300 mg/m^2 daily for 3 days and fludarabine 30 mg/m^2 daily for 3 days. The intent of chemotherapy is to enhance CAR T-cell activity.
* After the chemotherapy ends, the patients will have two days with no treatments and then receive an infusion of CAR T cells.
* The initial dose level will be 0.66x10^6 Anti-SLAMF7-CAR + T cells/kg of recipient bodyweight.
* The cell dose administered will be escalated for up to 4 doses until a maximum tolerated dose is determined.
* Following the T-cell infusion, there will be a mandatory 9-day minimum inpatient hospitalization to monitor for toxicity.
* Outpatient follow-up is planned for 2 weeks, and 1, 2, 3, 4, 6, 9, and 12 months after the CAR T-cell infusion. Afterwards, follow-up will be every six months up to at least 3 years after infusion.

ELIGIBILITY:
* INCLUSION CRITERIA - MULTIPLE MYELOMA:
* Signaling lymphocytic activation molecule F7 (SLAMF7) expression must be detected on malignant plasma cells from either bone marrow or a plasmacytoma by flow cytometry or immunohistochemistry. A specific quantitative level of SLAMF7 expression for eligibility is not specified, but patients with multiple myeloma cells that are negative for SLAMF7 by flow cytometry and immunohistochemistry will not be enrolled. These assays must be performed at the National Institutes of Health (NIH). It is not required that the specimen used for SLAMF7 determination comes from a sample that was obtained after the patient's most recent treatment. If paraffin embedded unstained samples of bone marrow involved with MM or a plasmacytoma are available, these can be shipped to the NIH for SLAMF7 staining, otherwise new biopsies will need to be performed for determination of SLAMF7 expression.
* SLAMF7 expression will need to be documented on the majority of malignant plasma cells by flow cytometry at the NIH at some time after the original chimeric antigen receptor (CAR)-SLAMF7 T-cell infusion in all patients undergoing a second CAR-SLAMF7 T-cell infusion on this clinical trial.
* Bone marrow plasma cells must make up less than or equal to 50% of total bone marrow cells based on a bone marrow biopsy performed within 24 days of the start of protocol treatment.
* Patients must have received at least 3 different prior treatment regimens for multiple myeloma (MM)
* Must have prior exposure to an immunomodulatory drug (IMiD) such as lenalidomide and a proteasome inhibitor
* Patients must have measurable MM as defined by at least one of the criteria below.

  * Serum M-protein greater or equal to 0.6 g/dL.
  * Urine M-protein greater or equal to 200 mg/24 h.
  * Serum free light chain (FLC) assay: involved FLC level greater or equal to 10 mg/dL (100 mg/L) provided serum FLC ratio is abnormal.
  * A biopsy-proven plasmacytoma at least 1.5 cm in largest dimension
  * Bone marrow core biopsy with 30% or more plasma cells

INCLUSION CRITERIA - OTHER:

* Greater than or equal to 18 years of age and less than or equal to age 73.
* Able to understand and sign the Informed Consent Document.
* Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0-2
* Patients of both sexes must be willing to practice birth control from the time of enrollment on this study and for four months after last day of receiving protocol treatment.
* Seronegative for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune-competence and thus are less responsive to the experimental treatment and more susceptible to its toxicities.)
* A patient with a negative blood polymerase chain reaction (PCR) test for hepatitis B deoxyribonucleic (DNA) test can be enrolled. If hepatitis B DNA (PCR) testing is not available, patients with a negative hepatitis B surface antigen and negative hepatitis B core antibody can be enrolled.
* Patients must be tested for the presence of Hepatitis C antigen by PCR and be hepatitis C virus (HCV) ribonucleic acid (RNA) negative in order to be eligible. Only if Hepatitis C PCR testing is not available in a timely manner, patients who are Hepatitis C antibody-negative can be enrolled.
* Absolute neutrophil count greater than or equal to 1000/mm^3 without the support of filgrastim or other growth factors within the previous 10 days.
* Platelet count greater than or equal to 55,000/mm^3 without transfusion support in the past 14 days.
* Hemoglobin greater than or equal to 8.0 g/dL.
* Less than 5% plasma cells in the peripheral blood leukocytes
* Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less or equal to 2.5 times the upper limit of the institutional normal.
* Serum creatinine less than or equal to 1.5 mg/dL.
* Total bilirubin less than or equal to 2.0 mg/dL, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dL.
* At least 14 days must have elapsed since any prior systemic therapy at the time the patient starts the cyclophosphamide and fludarabine conditioning regimen, and patients toxicities must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo or cytopenias).
* Because this protocol requires collection of autologous blood cells by leukapheresis in order to prepare CAR-SLAMF7 T cells, systemic anti-myeloma therapy including systemic corticosteroid steroid therapy of greater than 5 mg/day of prednisone or equivalent dose of another corticosteroid are not allowed within 14 days prior to the required leukapheresis.
* Normal cardiac ejection fraction (greater than or equal to 50% by echocardiography) and no evidence of hemodynamically significant pericardial effusion as determined by an echocardiogram.
* For patients with past participation in gene-therapy, cryopreserved peripheral blood mononuclear cells (PBMC) that have not been genetically engineered must be available.
* Patients receiving prior gene therapy outside of NIH will not be eligible. Patients who previously received CAR T-cell therapy at the National Cancer Institute (NCI) will be potentially eligible.

EXCLUSION CRITERIA:

* Patients who are receiving any other investigational agents.
* Patients on any anticoagulants except aspirin
* Patients that require urgent therapy due to tumor mass effects or spinal cord compression.
* Patients that have active hemolytic anemia.
* Patients with second malignancies in addition to multiple myeloma are not eligible if the second malignancy has required treatment within the past 3 years or is not in complete remission. There are two exceptions to this criterion: successfully treated non-metastatic basal cell or squamous cell skin carcinoma.
* Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant. Women of child bearing potential cannot have a positive pregnancy test. Women of childbearing potential are defined as all women except women who are post-menopausal or who have had a hysterectomy. Postmenopausal will be defined as women over the age of 55 who have not had a menstrual period in at least 1 year.
* Active systemic infections (defined as infections causing fevers or requiring anti-microbial treatment), active coagulation disorders or other major uncontrolled illnesses of the cardiovascular, respiratory, endocrine, renal, gastrointestinal, genitourinary, neurologic, psychiatric, or immune system, history of myocardial infarction, active cardiac arrhythmias, active obstructive or restrictive pulmonary disease.
* Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
* Systemic corticosteroid steroid therapy of greater than 5 mg/day of prednisone or equivalent dose of another corticosteroid (prednisone, dexamethasone, etc.) is not allowed within 14 days prior to either the required leukapheresis or within 14 days prior to CAR Tcell infusion (and at any time after the CAR T-cell infusion unless approved by the Principal Investigator or an Associate Investigator).
* History of severe immediate hypersensitivity reaction to any of the agents used in this study.
* Patient unwilling to undergo intensive care unit treatment including mechanical ventilation, cardiopulmonary resuscitation, vasoactive drugs, and hemodialysis.
* History of allogeneic stem cell transplantation
* Patients with current spinal cord compression (without intradural myeloma involvement.
* Patients who have a history (or current evidence) of cerebrospinal fluid multiple myeloma, or intradural central nervous system masses.
* Patients with active autoimmune skin diseases such as psoriasis or other active autoimmune diseases such as rheumatoid arthritis.
* Patients must not have required supplemental oxygen within the past month unless it was for a resolved infection.

Ages: 18 Years to 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2020-10-13 (Actual); Study Completion 2021-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James N Kochenderfer, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-C-0102.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3/13 participants enrolled on Level 2 (n=1) and Level 3 (n=2) were not treated,
Groups:
- LEVEL 1 - 0.66x10^6 Per Kilogram (kg): 0.66x10^6 Anti-Signaling lymphocytic activation molecule F7 (SLAMF7) - Chimeric antigen receptor (CAR) + T cells per kg of recipient bodyweight
- LEVEL 2 - 2.0x10^6 Per kg: 2.0x10^6 Anti-Signaling lymphocytic activation molecule F7 (SLAMF7) - Chimeric antigen receptor (CAR) + T cells per kg of recipient bodyweight
- LEVEL 3 - 6.0x10^6 Per kg: 6.0x10^6 Anti-Signaling lymphocytic activation molecule F7 (SLAMF7) - Chimeric antigen receptor (CAR) + T cells per kg of recipient bodyweight
- LEVEL 4 - 12.0x10^6 Per kg: 12.0x10^6 Chimeric antigen receptor (CAR) + T cells per kg of recipient bodyweight
Period: Overall Study
Arm/Group | LEVEL 1 - 0.66x10^6 Per Kilogram (kg) | LEVEL 2 - 2.0x10^6 Per kg | LEVEL 3 - 6.0x10^6 Per kg | LEVEL 4 - 12.0x10^6 Per kg
Started | 3 | 4 | 5 | 1
Completed | 3 | 3 | 3 | 1
Not Completed | 0 | 1 | 2 | 0
Not completed — Received anti-myeloma prescription (Rx) | 0 | 1 | 0 | 0
Not completed — No longer meets eligibility criteria | 0 | 0 | 1 | 0
Not completed — Started anti-cancer treatment | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: 3/13 participants not treated in Level 2 (n=1) and Level 5 (n=2) collected baseline data is reported in the table.
Groups:
- Total: Total of all reporting groups
Arm/Group | LEVEL 1 - 0.66x10^6 Per Kilogram (kg) | LEVEL 2 - 2.0x10^6 Per kg | LEVEL 3 - 6.0x10^6 Per kg | LEVEL 4 - 12.0x10^6 Per kg | Total
Number analyzed (Participants) | 3 | 4 | 5 | 1 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 5 | 1 | 12
  >=65 years | 0 | 1 | 0 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.33 (5.42) | 50.05 (11.9) | 53.61 (5.68) | 64.7 (0) | 54.83 (8.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3 | 0 | 6
  Male | 3 | 1 | 2 | 1 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 4 | 5 | 1 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 3 | 0 | 4
  White | 2 | 4 | 1 | 1 | 8
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 5 | 1 | 13
Number of Prior Lines of Therapy [Number; unit: prior therapy] — Population: Each row represents one participant.
  prior therapy
    Participant 1: number analyzed (Participants) | 1 | 0 | 0 | 0 | 1
    Participant 1 | 6 |  |  |  | 6
    Participant 2: number analyzed (Participants) | 1 | 0 | 0 | 0 | 1
    Participant 2 | 4 |  |  |  | 4
    Participant 3: number analyzed (Participants) | 1 | 0 | 0 | 0 | 1
    Participant 3 | 3 |  |  |  | 3
    Participant 4: number analyzed (Participants) | 0 | 1 | 0 | 0 | 1
    Participant 4 |  | 7 |  |  | 7
    Participant 5: number analyzed (Participants) | 0 | 1 | 0 | 0 | 1
    Participant 5 |  | 6 |  |  | 6
    Participant 6: number analyzed (Participants) | 0 | 1 | 0 | 0 | 1
    Participant 6 |  | 6 |  |  | 6
    Participant 7: number analyzed (Participants) | 0 | 0 | 1 | 0 | 1
    Participant 7 |  |  | 4 |  | 4
    Participant 8: number analyzed (Participants) | 0 | 0 | 1 | 0 | 1
    Participant 8 |  |  | 8 |  | 8
    Participant 9: number analyzed (Participants) | 0 | 0 | 1 | 0 | 1
    Participant 9 |  |  | 5 |  | 5
    Participant 10: number analyzed (Participants) | 0 | 0 | 0 | 1 | 1
    Participant 10 |  |  |  | 5 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Had Any Grade ≤2, and 3, 4 and 5 Adverse Events Following Administration of T Cells Expressing Anti- Signaling Lymphocytic Activation Molecule F7 (SLAMF7) Chimeric Antigen Receptor (CAR)
Description: Adverse Events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). Grade1 is mild, Grade 2 is moderate, Grade 3 is severe, Grade 4 is life-threatening or disabling, and Grade 5 is fatal.
Time Frame: Date treatment consent signed to date off study, approximately 3 months and 27 days for Level 1, 3 months and 18 days for Level 2, 5 months and 23 days for Level 3, and 1 month and 29 days for Level 4.
Population: 3/13 participants enrolled on Level 2 (n=1) and Level 3 (n=2) were not treated,
Measure: Count of Participants; unit: Participants
Arm/Group | LEVEL 1 - 0.66x10^6 Per Kilogram (kg) | LEVEL 2 - 2.0x10^6 Per kg | LEVEL 3 - 6.0x10^6 Per kg | LEVEL 4 - 12.0x10^6 Per kg
Number analyzed (Participants) | 3 | 3 | 3 | 1
Participants
  < Grade 2 | 0 | 0 | 1 | 0
  Grade 2 | 3 | 3 | 3 | 1
  Grade 3 | 3 | 3 | 3 | 1
  Grade 4 | 3 | 3 | 3 | 1
  Grade 5 | 0 | 0 | 0 | 0

2. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: as for outcome 1
Population: 3/13 participants enrolled on Level 2 (n=1) and Level 3 (n=2) were not treated,
Measure: Count of Participants; unit: Participants
Arm/Group | LEVEL 1 - 0.66x10^6 Per Kilogram (kg) | LEVEL 2 - 2.0x10^6 Per kg | LEVEL 3 - 6.0x10^6 Per kg | LEVEL 4 - 12.0x10^6 Per kg
Number analyzed (Participants) | 3 | 3 | 3 | 1
Participants | 3 | 3 | 3 | 1

3. Other Pre Specified Outcome: Number of Participants With a Response
Description: Response was assessed by the International Uniform Response Criteria for Multiple myeloma 2016 updated version. Complete Remission (CR) is negative immunofixation on the serum and urine, and disappearance of any soft tissue plasmacytomas. Very Good Partial Remission (VGPR) is serum and urine M-protein detectable by immunofixation but not on electrophoresis, or 90% or greater reduction in serum M-protein plus urine M-protein level <100mg per 24 h. Partial Remission (PR) is 50% or greater reduction of serum M-protein and 90% or greater reduction in 24-h urinary M-protein (or to less than 200mg per 24 h). Progressive Disease (PD) is serum M-component (minimum absolute increase of 0.5g/dL), or urine M-component (minimum absolute increase of 200mg/24h). Stable Disease (SD) is not meeting criteria for CR, VGPR, PR or progressive disease.
Time Frame: At two and five weeks for stable disease and partial remission, respectively, and up to 5 months and 23 days for progressive disease
Population: 3/13 participants enrolled on Level 2 (n=1) and Level 3 (n=2) were not treated. No weeks are necessary for PD.
Measure: Count of Participants; unit: Participants
Arm/Group | LEVEL 1 - 0.66x10^6 Per Kilogram (kg) | LEVEL 2 - 2.0x10^6 Per kg | LEVEL 3 - 6.0x10^6 Per kg | LEVEL 4 - 12.0x10^6 Per kg
Number analyzed (Participants) | 3 | 3 | 3 | 1
Participants
  Partial Remission at 5 Weeks | 0 | 1 | 0 | 0
  Stable Disease at 2 Weeks | 2 | 1 | 2 | 1
  Progressive Disease | 1 | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 3 months and 27 days for Level 1, 3 months and 18 days for Level 2, 5 months and 23 days for Level 3, and 1 month and 29 days for Level 4.
Arm/Group | LEVEL 1 - 0.66x10^6 Per Kilogram (kg) | LEVEL 2 - 2.0x10^6 Per kg | LEVEL 3 - 6.0x10^6 Per kg | LEVEL 4 - 12.0x10^6 Per kg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 1/3 | 1/1
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LEVEL 1 - 0.66x10^6 Per Kilogram (kg) (N=3) | LEVEL 2 - 2.0x10^6 Per kg (N=3) | LEVEL 3 - 6.0x10^6 Per kg (N=3) | LEVEL 4 - 12.0x10^6 Per kg (N=1)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LEVEL 1 - 0.66x10^6 Per Kilogram (kg) (N=3) | LEVEL 2 - 2.0x10^6 Per kg (N=3) | LEVEL 3 - 6.0x10^6 Per kg (N=3) | LEVEL 4 - 12.0x10^6 Per kg (N=1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (5) | 3 (8) | 3 (13) | 1 (8)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CPK increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 2 (3) | 1 (2)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (3) | 1 (1) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (9) | 1 (3)
Hypokalemia (Metabolism and nutrition disorders) | 2 (5) | 1 (4) | 0 (0) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 3 (7) | 1 (3)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, staph. Epidermidis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 3 (10) | 2 (5) | 3 (13) | 1 (7)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Actinic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 3 (11) | 3 (12) | 3 (10) | 1 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 2 (4) | 3 (8) | 1 (6)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 3 (24) | 3 (14) | 3 (10) | 1 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-14): https://cdn.clinicaltrials.gov/large-docs/56/NCT03958656/Prot_SAP_000.pdf
  • Informed Consent Form (2020-06-16): https://cdn.clinicaltrials.gov/large-docs/56/NCT03958656/ICF_001.pdf